CLINICAL TRIAL: NCT02310334
Title: The Impact of Real-Time Physiological Status Based Pacing Guidance on Physiological Strain for Exercising Humans
Brief Title: The Pacing (Guided Vs Unguided) Strategies Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Rumpler, Resesarch Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: HS47
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unguided Pacing Strategy (Experimental): Each participant will stay in the calorimeter (~24 hrs) on 2 different occasions. During the first visit, the participant will partake in an unguided exercise session.
  Interventions: Other: Guided Exercise Session
- Guided Pacing Strategy (Experimental): Each participant will stay in the calorimeter (~24 hrs) on 2 different occasions. During the second visit, the participant will partake in a guided exercise session.
  Interventions: Other: Unguided Exercise Session

INTERVENTIONS:
Other: Guided Exercise Session — Participants will be provided a pace based upon their current (estimated) physiological strain index (PSI) - a measure of thermal work strain, the time, and the distance completed already.
  Arms: Unguided Pacing Strategy
Other: Unguided Exercise Session — Participants will be instructed to complete 5 miles within 60 minutes and finish in as cool (lower body temperature) a state as possible.
  Arms: Guided Pacing Strategy

SUMMARY:
The objectives of this study are to demonstrate that real time physiological status monitoring and the use of optimization techniques during exercise can have a positive impact on physiological status, and to collect metabolic flexibility profiles of young fit adults during rest and exercise.

DETAILED DESCRIPTION:
This experiment aims to accomplish two goals: collect additional metabolic flexibility data with young fit adults in response to exercise; and demonstrate that automated pace guidance generated from real-time thermal-work strain monitoring and an optimized pacing policy will allow less stressful completion of a timed (60 minute) treadmill exercise of 5 miles. Each participant will undergo two treatments of first UNGUIDED followed by GUIDED exercise. The two exercise sessions will be conducted as part of a ~24 hour stay in an indirect calorimetry chamber.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Ages 18 to 29 at the beginning of the study
* Relatively fit can run 2 miles in under 16 minutes

Exclusion Criteria:

* History of Skin Sensitivity to Nickel
* Hypertension
* Alcoholism
* Diabetes
* Pregnant
* Age >29
* Cannot run 2 miles in less than 16 minutes
* No regular weekly exercise
* Difficulty Swallowing Food or Large Pills
* Diverticulitis
* Inflammatory Bowel Disease
* Peptic Ulcer Disease
* Crohn's Disease
* Ulcerative Colitis
* Previous Gastrointestinal Surgery
* Possible Nuclear Magnetic Resonance Scan
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* History or presence of kidney disease, liver disease, certain cancers, gastrointestinal, pancreatic, other metabolic diseases, or malabsorption syndromes
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (for at least 6 months prior to the start of the study)
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 12 months or who plan to initiate a weight loss program during the next 10 months
* Unable or unwilling to give informed consent or communicate with study staff.
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol
* Blood donation within the previous month

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Physiological Strain Index (PSI) | During 2-hour exercise session
  The PSI is an index that combines heart rate and core body temperatures with equal weights into an index from 0 to 10+. PSI will be calculated according to Moran et al. (1998) from measures of heart rate and core body temperature.

SECONDARY OUTCOMES:
Metabolic Flexibility | 24 hours
  O2 utilization and CO2 production will be analyzed during each calorimeter stay and used to measure metabolic rate indirectly.
Continuous Glucose Monitoring | 24 hours
  Continuous glucose monitoring will be used to examine the effects of the exercise regime on blood glucose.
Self Perception Scales | During 2-hour exercise session
  Self perception scales will be used that measure mood state, perceived exertion, thermal sensation, physical stresses and motivation.
Profile of Mood States (POMS) Questionnaire | During 2-hour exercise session
  The POMS is an inventory of subjective mood states (McNair, Lorr and Droppleman, 1992).
Thermal Sensation Scale | During 2-hour exercise session
  Two thermal sensation scales (original and modified) will be used to assess the thermal sensation of volunteers.
Perceived Exertion Scale | During 2-hour exercise session
  The Borg (1970) rating of perceived exertion (RPE) will be used.
Feeling Scale | During 2-hour exercise session
  The feeling scale will be used as an affective valence measure of exercise.
Motivation | During 2-hour exercise session
  Question will be asked to assess motivation during each exercise session.

CONTACTS AND LOCATIONS:
Overall Officials: William V Rumpler, PhD, Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States